CLINICAL TRIAL: NCT01302639
Title: Dietary Polyphenols as Modulators of Lipid Oxidation and Mitochondrial Function in Overweight Volunteers
Brief Title: Dietary Polyphenols and Lipid Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 10-03-032.7
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Obesity, Insulin Sensitivity, Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- EGCG and resveratrol (Experimental)
  Interventions: Dietary Supplement: Comparison of different combinations of polyphenols with respect to effects on fat oxidation
- EGCG, resveratrol and genistein (Experimental)
  Interventions: Dietary Supplement: Comparison of different combinations of polyphenols with respect to effects on fat oxidation
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Comparison of different combinations of polyphenols with respect to effects on fat oxidation

INTERVENTIONS:
Dietary Supplement: Comparison of different combinations of polyphenols with respect to effects on fat oxidation — EGCG, resveratol and genistein

SUMMARY:
There are strong indications that (combinations of) polyphenols may be attractive candidates in the prevention of the metabolic syndrome and diabetes through modulation of pathways of fatty acid metabolism and mitochondrial function. We hypothesize that the combination of specific polyphenols, with partly distinct mechanisms of action, may have physiologically significant effects on fat oxidation through additive or synergistic effects, thereby improving body composition, insulin sensitivity and preventing type 2 diabetes. The following objective will be addressed in the current study:

(1) to test short term (3 day) effects of combinations of polyphenols (supplements of EGCG either in combination with resveratrol or with resveratrol and genistein) to affect systemic lipolysis and fat oxidation during overnight fasted conditions and after ingestion of a high fat meal in overweight subjects

ELIGIBILITY:
Inclusion Criteria:

* overweight men and women (BMI≥25kg/m2- 29.9 kg/m2), aged 30-70 years, Caucasian, normal fasting glucose (< 6.1 mmol/L) and blood pressure (systolic blood pressure 100-140 mmHg, diastolic blood pressure 60-90 mmHg), weight stable in last 3 months (± 2kg). Exclusion criteria:

Exclusion Criteria:

* women lactating, pregnant or (post)menopausal, regular smokers, people with intensive fitness training, eg. athletes (≥ 3 per week ≥ 1 hour training), habitual consumption of green tea (more than 1 cup per day) or products containing green tea extract, total caffeine consumption > 300 mg/day, alcohol intake >20 g/day, any dietary vitamins or dietary supplements, diabetes mellitus (defined as FPG ≥ 7.0 mmol/l and/or 2hPG ≥ 11.1 mmol/l); serious pulmonary, cardiovascular, hepatic or renal disease : history of cardiovascular disease, all other relevant medical disorders that potentially interfere with this trial, current use of medication interfering with study intervention or interfering with study endpoints/hypotheses.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
postprandial fat oxidation | 3 days
  3 day supplementation of different combinations of polyphenols in a randomised crossover design in healthy overweight volunteers.
  At the end of each supplementation period, postprandial fat oxidation is measured

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Most J, Goossens GH, Jocken JW, Blaak EE. Short-term supplementation with a specific combination of dietary polyphenols increases energy expenditure and alters substrate metabolism in overweight subjects. Int J Obes (Lond). 2014 May;38(5):698-706. doi: 10.1038/ijo.2013.231. Epub 2013 Dec 9. PMID 24317366